CLINICAL TRIAL: NCT01658527
Title: Phase II Randomized Comparative Trial of TAK-700 (Orteronel) Versus Bicalutamide in Metastatic Prostate Cancer Patients Failing 1st Line Treatment With LHRH Agonists or Surgical Castration.
Brief Title: TAK-700 in Castration Resistant Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Pharmaceutical company has terminated orteronel (TAK-700) development for Prostate Cancer
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1211-GUCG-IG; 2012-002122-67 (EudraCT Number)
Record Dates: First submitted 2012-07-27; First posted 2012-08-07 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Cancer
Keywords: metastatic; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — orteronel; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orteronel, 300 mg twice daily (Experimental)
  Interventions: Drug: Orteronel
- Bicalutamide 50 mg per day (Active Comparator)
  Interventions: Drug: Bicalutamide

INTERVENTIONS:
Drug: Orteronel — Tak-700 will be administered until disease progression, diagnosis of a second malignancy, patient refusal to continue the treatment, excessive toxicity precluding further therapy according to protocol and /or according to the responsible physician.
  Upon progression, patient may stay on study medication until the initiation of a new therapy
  Other Names: TAK 700
  Arms: Orteronel, 300 mg twice daily
Drug: Bicalutamide — Bicalutamide will be given at the standard daily dose of 50 mg PO (per os). Bicalutamide will be maintained until disease progression diagnosis of a second malignancy, patient refusal to continue the treatment, excessive toxicity precluding further therapy according to protocol and /or according to the responsible physician.
  Arms: Bicalutamide 50 mg per day

SUMMARY:
The objective of this randomized phase II open label trial is to determine the anti-tumor activity of TAK-700 (Orteronel) as compared to bicalutamide in terms of clinical progression-free survival in prostate cancer patients who failed 1st line treatment with LHRH (luteinizing hormone-releasing hormone) agonists or surgical castration.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed diagnosis of prostate adenocarcinoma
* Metastatic disease in bone or other lesions documented by imaging. Abnormal 99mTc-bone scan imaging must be confirmed by Computed Tomography (CT) Scan or Magnetic resonance Imaging (MRI)
* Progressive disease following 1st line androgen deprivation therapy with LHRH (luteinizing hormone-releasing hormone) Agonists or surgical castration. Recommendations of Prostate Cancer Working Group 2 (PCWG2)
* WHO (World health organization) performance status ≤ 2
* Life expectancy > 12 weeks
* Adequate bone marrow function (Absolute neutrophil count (ANC) 1500/μL; platelets 100,000/μL)
* Castrate serum levels of testosterone (< 50 ng/dL)
* Adequate renal function: calculated creatinine clearance > 40 mL/minute
* Adequate hepatic function:

  * Bilirubin: total bilirubin 1.5 Upper limit of Normal (ULN)
  * Asparate aminotransferase (AST) and/or Alanine aminotransferase (ALT) ≤ 2.5 x ULN in the absence of liver metastases or ≤ 5 x ULN if liver metastases are present
* Patients of reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 4 months following the last study treatment. A highly effective method of birth control is defined as those that result in low failure rate (i.e. less than 1% per year) when used consistently and correctly
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP (International conference on Harmonization-Good Clinical Practices), and national/local regulations

Exclusion criteria

* Cardiac function:

  * Screening calculated ejection fraction (Multi Gated Acquisition Scan (MUGA) scan, or by echocardiogram) must be ≥ 50%
  * No history of myocardial infarction, unstable symptomatic ischemic heart disease, ongoing arrhythmias of Grade > 2 thromboembolic events (e.g., deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), or any other cardiac condition (e.g., pericardial effusion restrictive cardiomyopathy) within 6 months prior to first dose of study drug
  * Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed
  * Absence of New York Heart Association Class III or IV heart failure
  * Absence of Electrocardiogram (ECG) abnormalities of: Q-wave infarction, unless identified 6 or more months prior to screening and QTc interval > 470 msec
  * No uncontrolled hypertension despite appropriate medical therapy defined as blood pressure >160/90 mmHg at 2 separate measurements no more than 60 minutes apart during the Screening visit
* Prior radiotherapy but only for lymph nodes is allowed
* Prior or concomitant therapy:

  * No intake of narcotic analgesia for bone pain
  * No prior treatment with non-steroidal antiandrogens, within 6 months prior to randomization
  * No anticancer therapy or treatment with another investigational agent within the last 4 weeks prior to randomization
  * No prior therapy with TAK-700, ketoconazole, abiraterone, aminoglutethimide or MDV3100
  * Patients taking bisphosphonates or denosumab are eligible if they have received a stable dose for 4 weeks or more prior to randomization. (These treatments may then be continued on study)
* No known hypersensitivity to compounds related to TAK-700 or to TAK-700 excipients (refer to Investigator's brochure)
* No known gastrointestinal (GI) disease or GI procedure that could interfere with the GI absorption or tolerance of TAK-700, including difficulty swallowing tablets
* No prior history of adrenal insufficiency
* No prior history of malignancies other than prostate adenocarcinoma (except for basal cell or squamous cell carcinoma of the skin), or the patient has been free of malignancy for a period of 3 years prior to first dose of study drug
* No known active chronic hepatitis B or C, life-threatening illness unrelated to cancer, or any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with participation in this study
* No drug or alcohol abuse
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the trial is clinical progression free survival.
  The primary endpoint of the trial is clinical progression free survival. In this protocol, it is defined according to the recommendations of the "Prostate-Cancer clinical trials Working Group 2" and referred to as the "PCWG2" for the setting "delay/prevent" progression.

SECONDARY OUTCOMES:
RECIST (Response Evaluation Criteria In Solid Tumors) response in patients presenting with measurable disease
Time to PSA (Prostate specific antigen) progression and PSA change from baseline
Overall survival
Safety according to Common Terminology Criteria for Adverse Events, version 4.03
Pain (when an SAE (Serious Adverse Event)) or pain requiring initiation of narcotic analgesia
Skeletal related events, including requirement to initiate chemotherapy, radiotherapy, cord compression or requirement for surgery to the bone

CONTACTS AND LOCATIONS:
Overall Officials: Cora Sternberg, Principal Investigator — San Camillo Forlanini Hospitals, Rome, Italy; Bertrand Tombal, Study Chair — Cliniques Universitaires de St Luc, Brussels, Belgium
Locations (4):
- Belgium (4):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Cliniques Universitaires Saint-Luc, Brussels
  - AZ Groeninge Kortrijk - Campus Vercruysselaan, Kortrijck
  - CHU Dinant Godinne - UCL Namur, Yvoir